CLINICAL TRIAL: NCT00384618
Title: Effect of an Oxidative-Stress-Reducing Strategy Consisting of Pravastatin, Vitamin E and Homocysteine-Lowering on Carotid Intima-Media Thickness in Patients With Mild-to-Moderate Chronic Kidney Disease
Brief Title: Anti-Oxidant Therapy In Chronic Renal Insufficiency (ATIC) Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Medical Research Foundation, The Netherlands (Other); Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C97-1707
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2006-10-06 (Estimated); Status verified 2006-10

CONDITIONS: Chronic Kidney Disease
Keywords: Kidney, Antioxidants, Statin, Carotid IMT
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Pravastatin; Vitamin E

INTERVENTIONS:
Drug: pravastatin
Drug: vitamin E

SUMMARY:
The ATIC study is a randomised, double- blind, placebo-controlled trial in which the effects of oxidative stress-lowering treatment on vascular function and structure are studied in patients with chronic non-diabetic renal failure who are free from manifest arterial occlusive disease. Participants in the trial were randomised to active treatment consisting of add-on therapy with pravastatin, vitamin E and homocysteine-lowering therapy, or to placebo. Subjects not using angiotensin converting enzyme inhibitors (ACE-inhibitors) or angiotensin receptor blockers (ARBs) at inclusion were put on ACE-inhibitors for at least two weeks before the baseline measurement and randomisation. Those who were on ARBs continued their ARBs. We excluded individuals with diabetes mellitus (ADA criteria), active vasculitis, nephrotic syndrome (>3gr/24hr urine protein), renal transplantation, fasting total cholesterol > 7 mmol/L, cholesterol-lowering therapy within three months prior to inclusion or known ischemic cardiac, cerebrovascular or peripheral arterial disease. Ninety-three patients (out of 118 eligible patients) took part in the study and written informed consent was obtained from all participants.

DETAILED DESCRIPTION:
Background: Patients with mild-to-moderate renal failure have an increased risk of cardiovascular disease (CVD), which is not fully explained by the presence of classical cardiovascular risk factors. Oxidative stress has been proposed to play a major role in the development of CVD among renal failure patients. We investigated, in patients with mild-to-moderate chronic kidney disease (CKD), the effect of an oxidative-stress-lowering therapy with pravastatin, vitamin E and homocysteine-lowering on carotid intima-media thickness and endothelial function (two strong surrogate markers of cardiovascular risk), and renal function.

Methods: 93 patients with CKD (Cockcroft-Gault equation; mean: 41±17 ml / min per 1.73 m2) who were free of manifest arterial occlusive disease and diabetes mellitus were included in the Anti-oxidant Therapy In Chronic renal insufficiency (ATIC) study, a randomized, double-blind, placebo-controlled trial. The active treatment group received pravastatin 40 mg/day to which after 6 months vitamin E 300 mg/day was added and after another 6 months homocysteine-lowering therapy (folic acid 5 mg/day, pyridoxine 100 mg, vitamin B-12 1 mg/day). The placebo group received matching placebos at onset, and 6 and 12 months later. Blood pressure in both groups was managed according to a standard protocol to achieve a blood pressure of < 140/90 mmHg. Patients were followed up for two years. Measurements of common carotid artery intima-media thickness (CCA-IMT) and brachial artery endothelium-dependent, flow-mediated dilatation (BA-FMD) were performed at randomisation and after 6, 12 and 18 months. Plasma oxidized LDL (oxLDL) and plasma malondialdehyde (MDA) were measured as markers of oxidative stress at randomisation and after 6, 12, 18 and 24 months. We used generalized estimating equations (GEE) for data analysis.

ELIGIBILITY:
Inclusion Criteria:chronic

* kidney disease (clearence between 15-70ml/min)

Exclusion Criteria:

* diabetes mellitus (ADA criteria), active vasculitis, nephrotic syndrome (>3g protein/24h urine), renal transplantation, fasting total cholesterol > 7 mmol/L, cholesterol-lowering therapy within three months prior to inclusion or known ischaemic coronary, cerebrovascular or peripheral arterial disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-05; Study Completion 2005-08

PRIMARY OUTCOMES:
Common carotid artery intima media thickness
Brachial artery flow mediated vasodilatation

SECONDARY OUTCOMES:
Renal function

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Peter M ter Wee, MD, PhD, Study Director — Depratment of Nephrology, VU University Medical Center
Locations (1):
- VU University Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Result] Nanayakkara PW, Teerlink T, Stehouwer CD, Allajar D, Spijkerman A, Schalkwijk C, ter Wee PM, van Guldener C. Plasma asymmetric dimethylarginine (ADMA) concentration is independently associated with carotid intima-media thickness and plasma soluble vascular cell adhesion molecule-1 (sVCAM-1) concentration in patients with mild-to-moderate renal failure. Kidney Int. 2005 Nov;68(5):2230-6. doi: 10.1111/j.1523-1755.2005.00680.x. PMID 16221223
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745
- [Derived] Nanayakkara PW, Kiefte-de Jong JC, ter Wee PM, Stehouwer CD, van Ittersum FJ, Olthof MR, Teerlink T, Twisk JW, van Guldener C, Smulders YM. Randomized placebo-controlled trial assessing a treatment strategy consisting of pravastatin, vitamin E, and homocysteine lowering on plasma asymmetric dimethylarginine concentration in mild to moderate CKD. Am J Kidney Dis. 2009 Jan;53(1):41-50. doi: 10.1053/j.ajkd.2008.06.016. Epub 2008 Sep 11. PMID 18786751
- [Derived] Nanayakkara PW, van Guldener C, ter Wee PM, Scheffer PG, van Ittersum FJ, Twisk JW, Teerlink T, van Dorp W, Stehouwer CD. Effect of a treatment strategy consisting of pravastatin, vitamin E, and homocysteine lowering on carotid intima-media thickness, endothelial function, and renal function in patients with mild to moderate chronic kidney disease: results from the Anti-Oxidant Therapy in Chronic Renal Insufficiency (ATIC) Study. Arch Intern Med. 2007 Jun 25;167(12):1262-70. doi: 10.1001/archinte.167.12.1262. PMID 17592099